CLINICAL TRIAL: NCT00850941
Title: Radiation Therapy for Rising Prostate Specific Antigen (PSA) Post-prostatectomy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0254
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Prostate Cancer
Keywords: Registry; Research Database; Prostate cancer; Casodex; Flutamide; Goserelin Acetate; Leuprolide Acetate; Radiation; PSA; Post-prostatectomy; Radiation Therapy; Prostate Specific Antigen; Adenocarcinoma; Radical Prostatectomy; Bicalutamide; Zoladex; Lupron Depot; Tissue banking; Hormones
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — Surveys and Questionnaires; Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Leftover tissue from prostate surgery to be used for biomarker research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire: Prognostic factors and outcome for patients treated with radiation with curative intent for rising Prostate Specific Antigen (PSA) post-prostatectomy.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Information collection.
  Other Names: Registry; Survey; Quality of Life Survey

SUMMARY:
The goal of this clinical research study is to create a registry (research database) of clinical data about patients who receive radiation therapy, with or without hormone therapy, to treat prostate cancer that has come back after surgical removal of the prostate. This treatment is standard and the actual treatment is not part of this protocol.

The goal of this clinical research study is to create a registry (research database) of clinical data about patients who receive radiation therapy, with or without hormone therapy, to treat prostate cancer that has come back after surgical removal of the prostate. This treatment is standard and the actual treatment is not part of this protocol.

Researchers want to collect data and use this registry to learn about the long-term status of prostate cancer after these treatments.

This is an investigational study.

Up to 500 patients will take part in this study. All will be enrolled at MD Anderson, Spartanburg Regional Healthcare System, and/or MD Anderson Cancer Center Albuquerque.

Researchers want to collect data and use this registry to learn about the long-term status of prostate cancer after these treatments.

DETAILED DESCRIPTION:
Standard Treatment:

If you are found to be eligible and you choose to take part, you will be enrolled in this study. Study participants will be those who are receiving the standard radiation treatment for prostate cancer, which has come back after surgical removal of the prostate. If your PSA level is lower, you will receive radiation alone. If your PSA level is higher, you will receive hormone therapy in addition to radiation. You will sign a separate consent form that will describe these treatments and their risks in more detail. This study requires no other treatment. The main purpose of this study is data gathering through the use of questionnaires and tissue banking.

Follow-Up Tests

After your treatment (radiation with or without hormone therapy), you will receive routine follow-up care. The results of the following routine tests will be entered into the registry:

* After completing radiation, blood (about 1 tablespoon) will be drawn to check your PSA levels every 3 months for the first 2 years, every 6 months for the next 3 years, and every year from then on.
* If you receive hormone therapy, additional blood (about 1 tablespoon) will be drawn to check the levels of testosterone hormone. These blood tests to check your testosterone levels will be drawn at the same time as your PSA blood tests, until your testosterone levels are in the normal range.
* Every 6 months for the first 2 years after completing radiation, you will have a physical exam and a digital rectal exam. After that, the physical exam and digital rectal exam will be repeated every year from then on.

Information Collection:

While you are on study, on a long-term basis, researchers will collect information from your medical records about the status of the disease. This information will be entered into the registry. To identify you, the registry uses your medical record number instead of your name or other identifying information. The registry is password-protected to keep the data secure.

Length of Study Participation:

You will be on study for as long as you agree to keep taking part. If you go off study, your data will no longer be entered into the registry.

ELIGIBILITY:
Inclusion Criteria:

1. Adenocarcinoma of the prostate definitively treated by radical prostatectomy.
2. Patients must have no evidence of nodal or distant metastasis by clinical and radiologic staging to include bone scan and CT scan or MRI of the abdomen and pelvis. Patients with clinical or radiographic local recurrence are eligible. In patients with Gleason score less than or equal to 7 and PSA less than or equal to 1, CT or MRI of the abdomen is recommended but not required.
3. Rising PSA after prostatectomy defined as at least 2 consecutive rises. If total PSA < 0.2 ng/ml, surgical pathology must also show extracapsular extension, positive margins, or seminal vesicle involvement.
4. Total PSA < 5 ng/ml within 12 weeks prior to starting radiation or hormone therapy.
5. Patients with PSA greater than or equal to 0.5 ng/ml may have up to 3 months of an LHRH agonist and an anti-androgen immediately prior to enrollment.
6. All patient must have a serum testosterone of 150 ng/dl or greater documented prior to initiation of hormone therapy. Alternatively, patients without documentation of serum testosterone prior to initiation of hormone therapy should not have had any other prior hormone therapy within the 24 months preceding initiation of hormone therapy.

Exclusion Criteria:

1. Patients with pathologically positive pelvic lymph nodes at prostatectomy.
2. Patients with positive prostascint scans outside prostatic fossa.
3. Any chemotherapy, immunotherapy, biological therapy for cancer within 90 days of enrollment.
4. Hormone therapy (specifically LHRH agonist or antagonist, non-steroidal or steroidal antiandrogens) of more than 6 months duration at any time in the past for prostate cancer.
5. Contraindications to external beam radiation therapy to include previous pelvic radiation, inflammatory bowel disease or history of collagen vascular disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having a rising prostate-specific antigen (PSA) level after prostate was surgically removed, meaning prostate cancer return.
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2009-01-26 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Registry (research database) | Analyze data annually beginning once 100 patients have 1 year of follow-up; Anticipate annual enrollment of 100 patients.

SECONDARY OUTCOMES:
Quality of Life Assessment | At the 6 month, 1 year, 2 year, 3 year, 4 year, and 5 year follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Kuban, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Kaseman Presbyterian Hospital, Albuquerque, New Mexico
  - Spartanburg Regional Healthcare System, Spartanburg, South Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org